CLINICAL TRIAL: NCT03498066
Title: Assessment of βeta Blocker Interruption After Uncomplicated mYocardial Infarction on Safety and Symptomatic Cardiac Events Requiring Hospitalization: The AβYSS Study
Brief Title: Beta Blocker Interruption After Uncomplicated Myocardial Infarction
Acronym: AβYSS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Groupe Hospitalier Pitie-Salpetriere (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P150946J
Record Dates: First submitted 2018-03-21; First posted 2018-04-13 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: Myocardial Infarction
Keywords: Myocardial Infarction; Beta-Blockers; Stable Coronary Artery Disease
MeSH Terms: conditions — Myocardial Infarction | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Discontinuation of the Betablockers (βB) (Experimental): 1850 post-MI patients treated with chronic βB treatment will undergo withdrawal of their βB treatment..
  Interventions: Drug: Beta-blockers withdrawal
- Continuation of the Betablockers (βB) (Active Comparator): 1850 post-MI patients treated with chronic βB treatment will be continued under their usual βB treatment without modification.
  Interventions: Drug: Continuation of the Betablockers (βB) treatment

INTERVENTIONS:
Drug: Beta-blockers withdrawal — withdrawal of all type of betablockers
  Arms: Discontinuation of the Betablockers (βB)
Drug: Continuation of the Betablockers (βB) treatment — Use Betablockers treatment
  Arms: Continuation of the Betablockers (βB)

SUMMARY:
ABYSS is a national, multicenter, randomised, open label trial using the PROBE study design, that will evaluate the non-inferiority of the interruption of ΒB therapy after an uncomplicated MI after six months or more of follow-up compared to the continuation of βB evaluated by the primary endpoint or death, MI, Stroke and rehospitalization for others cardiovascular reasons.

DETAILED DESCRIPTION:
Despite the outstanding progress made in cardiac care over the last few years, cardiovascular diseases remain the leading cause of morbidity and mortality in developed countries.

After the initial clinical event, patients are considered to have a chronic disease which combined with the increasing actual life expectancy patients with CAD are a major source of expenses due to their life-long treatment and follow-up.

ΒB are prescribed during the initial hospitalisation for MI and in the post-MI phase. European (European Society of Cardiology, ESC) and American (ACC/AHA) guidelines initially gave βB therapy a class I recommendation for MI or acute coronary syndrome (ACS) for the first year of treatment and extended such recommendation without solid data up to 3 years after MI , . However, there has been no recent clinical trial to evaluate safety and efficacy of long term ΒB therapy in the contemporary therapeutic era. Taking such lack of evidence in account and acknowledging that clinical practice has changed, the latest ESC STEMI (2014) and NSTEMI (2015) Guidelines degraded the recommendation for the use of ΒB in post MI patients (Class IIa B) during the hospitalization period and they question the validity of its use after the initial stabilization phase. This was confirmed in the 2017 STEMI Guidelines.

The primary objective of the ABYSS trial is to demonstrate the non-inferiority of the interruption of ΒB therapy after an uncomplicated MI after six months or more of follow-up compared to the continuation of βB evaluated by the primary endpoint.

The primary endpoint of the study will be evaluated, with one-year minimum follow-up, and will be the composite of Major Adverse Cardiovascular Events (MACE) measured at the longest follow-up including:

* All-cause death
* Stroke
* Myocardial infarction Hospitalisation for other cardiovascular (CV) reason.

It is expected that the interruption of βB therapy will not alter the prognosis of patients and improve safety and quality of life of patients and considerably reduce healthcare direct or indirect costs.

ELIGIBILITY:
Inclusion criteria

Subjects meeting all of the following criteria will be considered for enrolment into the study:

1. Male or female +/=18 years of age
2. Current treatment with βB whatever the drug or the dose used
3. Prior acute myocardial infarction 6 months or more before randomisation defined either by:

   AβYSS protocol, version 3.0 of 25/05/2021 Page 32 / 65
   * An episode of ST elevation MI with ST segment elevation (STEMI) and/or the presence of Q wave (Type I MI)
   * an episode of Non ST Elevation MI (NSTEMI) with preferably at least one of the followings:

     * i) a documented hypokinetic or akinetic segment on echo or any other imaging technique
     * ii) segmental hypoperfusion Thallium or any other imaging technique
     * iii) segmental aspect of necrosis on MRI
   * An episode of silent MI discovered on ECG or Cardiac Imaging. Importantly = The mention of an MI on a report is enough to be considered as a prior MI and it is not necessary to retrieve the source document and/or documentation of this prior MI .
4. Patient affiliated to Social Security
5. Informed consent obtained in writing at enrolment into the study

Exclusion Criteria:

* Subjects presenting with any of the following will not be included in the study:

  1. Uncontrolled arterial hypertension according to investigator decision
  2. Prior episode of heart failure in the past two years of follow-up and/or low left ventricular ejection fraction <40% requiring the use of βB;
  3. New ACS (in the past 6 months) including UA/NSTEMI and STEMI;
  4. Persistent angina or ischemia (>10% viable myocardium) requiring the use of βB;
  5. Prior episode of ventricular or supraventricular arrhythmia in the past year of follow-up requiring the use of ΒB;
  6. Treatment with other investigational agents or devices within the previous 30 days, or previous enrolment in this trial.
  7. Pregnant Women or breast feeding women
  8. Patient under legal protection (protection of the court, or in curatorship or guardianship).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3700 (Actual)
Dates: Start 2018-08-29 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
The composite of Major Adverse Cardiovascular Events (MACE) | Through study completion, with a minimum of 1 year
  Will be evaluated with one-year minimum follow-up and will be the composite of Major Adverse Cardiovascular Events (MACE) including:
  * All-cause death
  * Myocardial infarction (MI)
  * Stroke
  * Hospitalisation for any cardiovascular (CV) reason.

SECONDARY OUTCOMES:
Quality of life | Through study completion, with a minimum of 1 year
  will be evaluated by the questionnaire EQ5D-5L Score (0 to 1) and EQ5D-5L Scale (0 to 100) with higher scores indicating a better quality of Life.

OTHER OUTCOMES:
Anxiety and Depression | Through study completion, with a minimum of 1 year
  will be evaluated by using the HADS questionnaire to detect the presence of depression and anxiety ( there is no score; this will be determined by the response selected by the patient with "no" = no discomfort to "a lot" = significant discomfort
Erection Dysfunction | Through study completion, with a minimum of 1 year
  A precise evaluation of Erectile dysfunction will be proposed to male patients using an internationally validated questionnaire IIEF (International Index of Erectile Function) in French with 5 questions whose answer is graded from 0 to 5 per question
Libido | Through study completion, with a minimum of 1 year
  An evaluation of lack of sex drive will be evaluated by answering the following questions about the sexuality of the patient The frequency and degree of sex drive (self evaluation)
Exercise Capacity | Through study completion, with a minimum of 1 year
  will be evaluated by answering the following simple questions :
  * The weekly physical activity and the sport practiced
  * Participation in competitions or not additionally, the recording the results of stress tests when available
  * Pre- and post - inclusion stress/ Strain test data
Side effects | Through study completion, with a minimum of 1 year
  will be evaluated by answering the following questions: Presence of Blury Vision, Sensation of cold hands and feets, Insomnia and palpitations

CONTACTS AND LOCATIONS:
Overall Officials: Johanne SILVAIN, MD-PhD, Study Chair — APHP / Institut de Cardiologie, Pitié-Salpêtrière Hospital, Paris (APHP) / ACTION Study Group / Sorbonne Université Paris-France
Locations (1):
- Institut de Cardiologie - USIC - Hôpital Pitié-Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available

REFERENCES:
- [Result] Silvain J, Cayla G, Ferrari E, Range G, Puymirat E, Delarche N, Collet JP, Dumaine R, Slama M, Payot L, Kasty ME, Aacha K, Vicaut E, Montalescot G; ABYSS investigators of the ACTION Study Group,. betaeta blocker interruption after uncomplicated myocardial infarction: rationale and design of the randomized ABYSS trial. Am Heart J. 2023 Apr;258:168-176. doi: 10.1016/j.ahj.2023.01.014. Epub 2023 Jan 20. PMID 36682596
- [Derived] Silvain J, Cayla G, Ferrari E, Range G, Puymirat E, Delarche N, Guedeney P, Cuisset T, Ivanes F, Lhermusier T, Petroni T, Lemesle G, Bresoles F, Labeque JN, Pommier T, Dillinger JG, Leclercq F, Boccara F, Lim P, Besseyre des Horts T, Fourme T, Jourda F, Furber A, Lattuca B, Redjimi N, Thuaire C, Deharo P, Procopi N, Dumaine R, Slama M, Payot L, El Kasty M, Aacha K, Diallo A, Vicaut E, Montalescot G; ABYSS Investigators of the ACTION Study Group. Beta-Blocker Interruption or Continuation after Myocardial Infarction. N Engl J Med. 2024 Oct 10;391(14):1277-1286. doi: 10.1056/NEJMoa2404204. Epub 2024 Aug 30. PMID 39213187
- [Derived] Granger CB, Pocock SJ, Gersh BJ. The need for new clinical trials of old cardiovascular drugs. Nat Rev Cardiol. 2023 Feb;20(2):71-72. doi: 10.1038/s41569-022-00819-1. No abstract available. PMID 36526898